CLINICAL TRIAL: NCT00371449
Title: Speech-in-Noise Measures as a Predictor of Hearing Aid Outcomes
Brief Title: Predicting Success With Hearing Aids
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: C4352-R
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hearing Loss; Presbycusis
Keywords: hearing loss; hearing aids
MeSH Terms: conditions — Hearing Loss; Presbycusis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hearing aid users: hearing aid users

SUMMARY:
The primary complaint of individuals with hearing loss is difficulty understanding speech in the presence of background noise. Although hearing aids help individuals understand speech in background noise better, there is a high rate of hearing aid rejection in part due to continued difficulty understanding speech in complex listening situations. The results of this study may demonstrate that speech-in-noise test results can be a predictor of hearing aid success. The results of this study also may lead to further studies that can evaluate interventions to improve hearing aid success for individuals who are identified as unsuccessful hearing aid users.

DETAILED DESCRIPTION:
As numerous studies have reported, the most common complaint that individuals with sensorineural hearing loss have about their hearing is that they can hear speech but they cannot understand speech, especially in background noise. For this type of hearing loss and most other types of hearing losses, hearing aids are the intervention of choice. The majority of individuals who receive hearing aids are successful hearing-aid users in that both subjectively and objectively they function better with their hearing aids than without hearing aids. Other individuals are unsuccessful hearing-aid users because for a variety of reasons their perception is that the hearing aids do not enable them to function better. Two studies (Popelka et al., 1998; Kockchin, 2000) indicate that about 25% of individuals who receive hearing aids can be considered unsuccessful hearing-aid users. If potentially (un)successful hearing-aid users can be identified, then audiologic rehabilitation programs can be designed for use with potentially successful hearing-aid users and more extensive audiologic rehabilitation programs can be designed for use with those individuals who are potentially unsuccessful hearing-aid users.

Data from a recent series of studies by N b lek and her colleagues (1991, 2004) indicate that successful and unsuccessful hearing-aids users can be predicted based on their performance on a subjective speech-in-noise task in which a most comfortable listening level is established for a travelogue story and the level of a multitalker babble is established that permits following the travelogue. The difference between these two levels is the acceptable noise level (ANL). Based on the ANL data, N b lek et al. (2006) report with 85% confidence those individuals who are successful hearing-aid users and those who are unsuccessful hearing-aid users. One premise of this proposal is that the ANL is in fact an estimate in the subjective realm of the signal-to-noise (S/N) at which the listener is comfortable listening to a speech signal in background noise.

Recently in our laboratory the words-in-noise (WIN) test was developed that involves the presentation of words in multitalker babble at signal-to-babble (S/B) ratios from 24- to 0-dB in 4-dB decrements. The 50% point on the function is calculated with the Spearman-K rber equation. This objective instrument provides an average 8-dB separation in recognition performances between listeners with normal hearing and listeners with hearing loss. The 50% points for the listeners with normal hearing are 0- and 6-dB S/B, whereas the 50% points for the listeners with hearing loss are 8- and 16-dB S/B. Thus, not only is the WIN very sensitive to the effects of hearing loss on speech understanding, but the WIN provides a range of performances by listeners with hearing loss.

The proposed study is designed to answer the following two key questions:

1. What is the relationship between ANL performance (subjective paradigm) and WIN performance (objective paradigm) in both unaided and aided conditions?
2. How well do the ANL and WIN scores predict subjective hearing-aid outcome domains (use, satisfaction, benefit, and global)?

In addition, the study design enables multiple comparisons to be made among several of the study variables and among many traditional variables such as age, pure-tone thresholds, and word-recognition abilities in quiet.

Future goals beyond this proposal involve the development (1) of systematic protocols to select amplification devices or specific features for amplification based on WIN or ANL performance, and (2) of audiologic rehabilitation programs that can be administered quickly and effectively (depending on the category of hearing-aid success that was determined from performances on the WIN or ANL) to veterans who are receiving hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* adult onset of hearing loss,
* symmetrical, sensorineural hearing loss,
* no more than 60 dB HL hearing loss measured via an average of air conduction thresholds at .5, 1, and 2 kHz in each ear, and
* use of binaural hearing aids of the same make and model for each ear
* at least 3 months of hearing aid use.

Exclusion Criteria:

* enrollment in group audiologic rehabilitation classes,
* currently using an FM system,
* inability to read and write American English, and
* signs of middle ear or retrocochlear pathology.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults with sensorineural hearing loss
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- James H. Quillen VA Medical Center, Mountain Home, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hearing-Aid Users: Individuals who wore hearing aids for > 3 months and at their current setting for at least 1 month
Period: Overall Study
Arm/Group | Hearing-Aid Users
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hearing Aid Users
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 120
degree of hearing loss [Mean (Standard Deviation); unit: dB HL] | 36.3 (10.8)
unaided Words-In-Noise Test [Mean (Standard Deviation); unit: dB S/N] | 14.4 (4.5)
unaided Acceptable Noise Level test [Mean (Standard Deviation); unit: dB] | 15.5 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Words-in-noise Test
Description: The WIN consists of two lists of 35 Northwestern University Auditory Test No. 6 words (NU-6; Tillman and Carhart, 1966) presented in a 6-talker babble at 7 SNRs ranging from 24- to 0-dB in 4-dB decrements. Thus for each list, five unique words spoken by a female talker are presented at each SNR with the level of the babble fixed (Department of Veterans Affairs, 2006). The SNR at which the 50% point occurs is calculated with the Spearman-Kärber equation (Finney, 1952). Normal performance on the WIN is between 0 and 6-dB S/N.
Time Frame: aided (after wearing hearing aids for at least 3 months)
Measure: Mean (Standard Deviation); unit: dB S/N
Groups:
- Group 1: hearing aid users
Arm/Group | Group 1
Number analyzed (Participants) | 120
dB S/N | 12.6 (3.7)

2. Secondary Outcome: Acceptable Noise Level Test
Description: The ANL consists of a speech signal and a competing noise signal. The speech signal is a continuous monologue (Arizona Travelogue) by a male talker and the competing noise signal is the 12-talker babble from the Speech in Noise (SPIN) test (Kalikow et al, 1977). The speech and babble stimuli are recorded on separate channels on a compact disc (CD; Cosmos, Inc.). The task of the listener was to adjust the level of the travelogue to the most comfortable level (MCL) and then to adjust the level of the babble to the level the listener is willing "to put up with" and still follow the travelogue, or to the background noise level (BNL). The ANL (in dB) is the difference between the MCL and BNL.
Time Frame: aided (after wearing hearing aids for at least 3 months)
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Hearing-aid Users: hearing aid users
Arm/Group | Hearing-aid Users
Number analyzed (Participants) | 120
dB | 13.5 (6.8)

3. Secondary Outcome: International Outcomes Inventory for Hearing Aids (IOI-HA)
Description: Overall/general hearing-aid outcome measure. Range in scores are 7-35 with higher scores representing better outcomes.
Time Frame: aided (after wearing hearing aids for at least 3 months)
Measure: Mean (Standard Deviation); unit: units on a scale (points)
Arm/Group | Hearing Aid Users
Number analyzed (Participants) | 120
units on a scale (points) | 28.9 (3.8)

4. Secondary Outcome: Measure of Audiologic Rehabilitation Self-Efficacy for Hearing Aids (MARS-HA)
Description: Measures hearing-aid self-efficacy over four subscales (basic handling, advanced handling, adjustment, and aided listening). Subscale scores are averaged to produce a total self-efficacy scores that can range from 0 (low self-efficacy) to 100 (high self-efficacy).
Time Frame: aided (after wearing hearing aids for at least 3 months)
Measure: Mean (Standard Deviation); unit: % level of self-efficacy
Arm/Group | Hearing Aid Users
Number analyzed (Participants) | 120
% level of self-efficacy | 84.7 (9.4)

5. Secondary Outcome: Satisfaction With Amplification in Daily Life (SADL)
Description: Measures how satisfied listeners are with their current hearing aids. Total scale scores are computed by averaging the subscale (positive effect, negative features, personal image, and service & delivery) scores that range from 1 (no satisfaction) to 7 (high satisfaction).
Time Frame: aided (after wearing hearing aids for at least 3 months)
Measure: Mean (Standard Deviation); unit: units on a scale (points)
Arm/Group | Hearing Aid Users
Number analyzed (Participants) | 120
units on a scale (points) | 5.4 (0.7)

6. Secondary Outcome: Speech Spatial and Qualities of Hearing Scale (SSQ)
Description: The SSQ measures hearing abilities related to speech, spatial perception, and quality of sound using a 1-10 scale. Items are averaged across the test. Higher scores indicate better outcomes.
Time Frame: aided (after wearing hearing aids for at least 3 months)
Measure: Mean (Standard Deviation); unit: units on a scale (points)
Arm/Group | Hearing Aid Users
Number analyzed (Participants) | 120
units on a scale (points) | 7.2 (1.4)

ADVERSE EVENTS:
Arm/Group | Hearing-aid Users
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No